CLINICAL TRIAL: NCT02804776
Title: PROGRESS: PRe-Operative Gefitinib in Resectable EGFR Mutation Positive Lung Cancer With Sector Sequencing for Biomarker Discovery
Brief Title: PRe-Operative Gefitinib in Resectable EGFR Mutation Positive Lung Cancer With Sector Sequencing for Biomarker Discovery
Acronym: PROGRESS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Centre, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ECRU-LUNG-2013
Record Dates: First submitted 2016-06-14; First posted 2016-06-17 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Gefitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gefitinib (Experimental): Gefitinib 250mg oral daily will be given for 4 weeks prior to surgery
  Interventions: Drug: Gefitinib

INTERVENTIONS:
Drug: Gefitinib — 250mg oral daily for 4 weeks
  Other Names: Iressa

SUMMARY:
This is a pharmacodynamic study to evaluate the effect of gefitinib as induction therapy for patients who have resectable, Epidermal growth factor receptor (EGFR) sensitizing mutation lung cancer.

DETAILED DESCRIPTION:
Selected patients will receive 4 weeks of gefitinib before surgery. A Positron Emission Tomography - Computed Tomography (PET- CT) will be performed before and after gefitinib to assess the response. Circulating tumour cells (CTCs) and plasma Deoxyribonucleic acid (DNA) will be acquired at baseline, 2 weeks and 4 weeks after gefitinib treatment. Resected tumor will be sectored in details to study the spatial heterogeneity.

ELIGIBILITY:
Inclusion Criteria:

* EGFR mutation positive Non-Small Cell lung cancer (NSCLC) (regardless of smoking status), or control group may encompass other molecular subtypes of lung cancer e.g. anaplastic lymphoma kinase (ALK) and Kirsten rat sarcoma viral oncogene homolog (KRAS).
* All early stage patients with NSCLC who are deemed surgically resectable.
* All patients must have histologically proven NSCLC, with known EGFR mutation
* Patients should be fit for either lobectomy/ pneumonectomy with or without lymph node sampling.
* Primary tumour should be at least 2 cm in size (Tumor stage 1b).
* Willing to provide informed consent.

Exclusion Criteria:

* Known severe hypersensitivity to gefitinib or any of the excipients of this product
* Any serious concomitant systemic disorder that, in the opinion of the investigator, would compromise the patient's ability to complete the study.
* Interstitial lung disease (ILD) or pulmonary fibrosis; impaired pulmonary function (e.g. FEV1 <40% predicted value, artery blood gas PaO2<60mmHg)
* Patients with prior exposure to agents directed at the Human epidermal receptor (HER) axis (e.g. erlotinib, gefitinib, cetuximab, trastuzumab).
* Patients with prior exposure to chemotherapy, irradiation or systemic anti-cancer therapy (e.g. monoclonal antibody therapy) for lung cancer.
* Any unstable systemic disease (including active infection, uncontrolled hypertension, unstable angina, congestive heart failure, myocardial infarction within six months, serious cardiac arrhythmia requiring medication, hepatic, renal, or metabolic disease).
* Evidence of any other disease, neurological or metabolic dysfunction, physical examination or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the subject at high risk for treatment-related complications.
* Patient who has serious active infection.
* Patients who harbouring exon 20 T(Threonine)790M (Methionine) mutation.
* Pregnancy or breast feeding.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-01-27 (Actual); Primary Completion 2018-02-21 (Actual); Study Completion 2018-02-21 (Actual)

PRIMARY OUTCOMES:
EGFR TKI sensitivity biomarkers determination | 4 to 6 weeks
  Determine EGFR tyrosine kinase inhibitor (TKI) sensitivity biomarkers in responders vs non responders, as categorized by either Response Evaluation Criteria In Solid Tumors (RECIST) stable disease (SD) vs Partial response (PR) or median percentage tumour shrinkage

SECONDARY OUTCOMES:
Response rates after 4 weeks of neoadjuvant gefitinib | 4 to 6 weeks
  To determine response rates after 4 weeks of neoadjuvant gefitinib as evaluated by RECIST 1.1

OTHER OUTCOMES:
Clonal heterogeneity using whole exome and RNA-sequencing of tumour sectors as well as resected lymph nodes | 4 to 6 weeks
Clonal heterogeneity recapitulation through CTC, plasma DNA and functional imaging | 4 to 6 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Daniel SW Tan, Principal Investigator — National Cancer Centre, Singapore
Locations (1):
- National Cancer Centre, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No